CLINICAL TRIAL: NCT06337188
Title: Adaptive and Individualized AAC Phase II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Altec Inc. (Industry)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAC PhII
Record Dates: First submitted 2024-03-18; First posted 2024-03-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Communication Disorders
MeSH Terms: conditions — Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental and Generic Communication Interfaces for AAC (Experimental): Each participant receives both Experimental and Generic AAC systems to communicate - in that order.
  Interventions: Device: Experimental AAC; Device: Generic AAC

INTERVENTIONS:
Device: Experimental AAC — Participant receives an AAC system comprising 2 wearable sensors for movement-mediated cursor control and muscle activity mediated cursor selection that is integrated with an adaptive and individualized keyboard to test communication performance.
Device: Generic AAC — Participant receives an AAC system that is similar to that used to satisfy their normal daily communication needs such as an eye-tracking device with a generic AAC keyboard to test communication.

SUMMARY:
The overall objective of this study is to develop an Augmentative and Alternative Communication (AAC) system that is effective in delivering a person-centric communication device that will provide a versatile access method that can automatically learn and adapt to the user's physical abilities by creating a personalized, comprehensive keyboard interface for communication, not otherwise available to people in need of alternative communication.

DETAILED DESCRIPTION:
The investigators propose an AAC device comprising a versatile access method that automatically learns and customizes a keyboard interface to the residual motor function of the individual. The team comprising scientists, speech researchers and clinicians is developing a prototype AAC system comprising versatile access method and personalized, comprehensive communication software. This will be achieved by developing hardware to support streamlined access across multiple points on the body, designing automated algorithms to rapidly create an expanded AAC interface, inclusive of letters, numbers, symbols, emojis, and word completion options, that is personalized based on the residual motor function of user-specific access points, creating software for point-of-care use of the access technology and interface, and evaluating the resulting AAC system for communication efficacy in individuals with severe motor impairments. The milestone will be to demonstrate that our AAC system improves Information Transfer Rate (ITR) and user experience over conventional AAC devices. The final AAC deliverable will be easily integrated with existing AAC tablets and mobile devices to provide those in need of alternative communication methods with an automatically customized, efficient, and intuitive solution to restore communication access in their daily lives. The project's involvement of human subjects for the purpose of research is primarily focused on testing our AAC system for usability, improved performance, acceptance, and perceived benefit among individuals with severe motor impairments.

ELIGIBILITY:
Inclusion Criteria:

* Adults or Children; age greater than or equal to 6 y.o.
* Male or female
* Able to (a) spell, (b) follow 2-3 step directions, (c) read 40 point text
* Have complex communication needs representing a broad spectrum of developmental and acquired severe motor impairments resulting from high spinal cord injury (SCI), chronic Guillain-Barre syndrome, brain stem stroke, cerebral palsy (CP), locked-in syndrome, among others.
* Requires the use of an alternative access strategy to communicate and/or use technology that has been clinically prescribed and manually optimized following current clinical standards.
* Sufficient control and voluntary muscle activation on either the head, hand, or foot (on the basis of clinical evaluation by clinical collaborators at University of Nebraska Medical Center) to use the proposed wearable AAC system for the purpose of this study.
* Sufficient stamina and developmental maturity (on the basis of clinical evaluation by clinical collaborators at University of Nebraska Medical Center) to attend to the approximately 1-2 hour protocols outlined in Aims 2 and 3 without excess fatigue or distraction.
* Availability for at least 5 testing sessions over the study period.
* No medical or safety restrictions of active head, hand, or foot movement (as determined by clinical collaborators at University of Nebraska Medical Center).
* Clinical evidence of preserved cognition by a score of 0 or 1 on NIHSS Consciousness and Communication item.
* Ability to voluntarily blink eyes or raise eyebrows on command (for head selection) or contract fingers/hand grasp (for hand selection) or rotate foot (for foot selection).
* Able to provide written, informed consent or an accompanying communication partner or parent/guardian (for individuals under 18 y.o) to provide written, informed consent/assent to participate in the study.
* Able to speak and follow directions in English.

Exclusion Criteria:

* Non-English speaker.
* Inability to follow simple instructions in English.
* Medical history of musculoskeletal conditions (arthritis, spondylosis, etc.) that causes pain on head, hand, or foot movement.
* Restricted active or passive rotation of head and neck resulting from unstable vertebral, spinal cord, or nerve roots that places the subject at risk for execution of the protocol.
* Medical history of cardiac or respiratory complications, or similar disorders that would severely reduce stamina and/or place the subject at risk for conducting the different motor activities.
* Unable to provide informed assent/consent in English.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Tele-healthcare Satisfaction Questionnaire - Wearable Technology (TSQ-WT) | 1 year
  Measures quantitative ratings on the TSQ-WT scale from a minimum rating of 0 to a maximum rating of 4, where the higher value means a better outcome.
Information Transfer Rate | 1 year
  Measures the speed in meters/second of accurately moving a cursor to a specified target on a computer screen.
National Aeronautics and Space Administration (NASA) Task Load Index | 1 year
  Measures qualitative ratings that are rated on an interval scale ranging from low (1) to high (100) of perceived user demand, performance, effort, and frustration.

SECONDARY OUTCOMES:
Character-to-character Movement Time | 1 year
  Measures the duration in seconds required to move a cursor to a specified target on a computer screen.
Path Efficiency | 1 year
  Measures the ratio of an ideal cursor path between targets to the actual path traveled.
Frequency of Selecting Word Completion Options | 1 year
  Measures the number of times per session a predicted word is chosen in place of spelling out the individual letters of the word.
Number of Written Disfluencies | 1 year
  Measures the number of times per session a target is substituted, inserted, or deleted as well as the number of pauses between target selections.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca De Luca, M.S., Principal Investigator — Altec Inc.
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No